CLINICAL TRIAL: NCT05585359
Title: Effect of Injectable Platelet Rich Fibrin Augmented With Vitamin C Compared to Injectable Platelet Rich Fibrin Alone on Healing of Necrotic Mature Single Rooted Teeth With Chronic Peri-apical Periodontitis Following Regenerative Endodontics (A Randomized Controlled Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wesam Osama Hassan Soliman, Assistant lecturer at Misr University for Science and Technology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5-6-1
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Periapical Periodontitis
Keywords: iprf; iprf with AA; periapical lesion
MeSH Terms: conditions — Periapical Periodontitis | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Parallel Randomized controlled blinding trail
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator will not be blinded due to the natural of the intervention and control which require blood withdrawal from the patient or to be mixed with the Vitamin C.
  * The patients and the outcome assessors are blinded to the intervention.
  * The patients will not be informed which technique of treatment will be used.
  * Data analyst will be blinded, he/she will receive data excel sheets with group A and group B
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable platelet rich fibrin with Vitamin C (Experimental): Injectable platelet rich fibrin: 10-mL sample of whole venous blood will be drawn from the patient's forearm and transferred into two plain plastic test tubes without an anticoagulant and will centrifuge immediately at 700 rpm for 3 minutes (60×g) . After centrifugation, the upper yellow fluid liquid (i-PRF) will be collected as close as possible to the layer of red cells the will be mixed with 250 micromole of Vitamin C.
  Interventions: Other: injectable platelet rich fibrin augmented with Vitamin C
- Injectable platelet rich fibrin alone (Active Comparator): injectable platelet rich fibrin: 10-mL sample of whole venous blood will be drawn from the patient's forearm and transferred into two plain plastic test tubes without an anticoagulant and will centrifuge immediately at 700 rpm for 3 minutes (60×g) . After centrifugation, the upper yellow fluid liquid (i-PRF) will be collected as close as possible to the layer of red cells
  Interventions: Other: injectable platelet rich fibrin augmented with Vitamin C

INTERVENTIONS:
Other: injectable platelet rich fibrin augmented with Vitamin C — According to the amount of the injectable platelet rich fibrin that will be obtained after the centrifugation of blood, the amount of Vitamin C will be calculated to be; for each 1 ml of injectable platelet rich fibrin, 250 μg of Vitamin C will be mixed with the i-PRF and injected inside the canals using a plastic syringe with a 25-gauge needle that was placed 1mm short of the working length and will be withdrawn gradually while injecting till reaching the canal orifice

SUMMARY:
The purpose of the study is to investigate the effect of injectable platelet rich fibrin augmented with Vitamin C (ascorbic acid) in healing of chronic peri-apical lesion, by assessing it radiographically 2dimensionally and 3 dimensionally

DETAILED DESCRIPTION:
all patients will be informed about the study through informed constant that will describe the natural of the study beside the potential risks of it. After accurate diagnosis clinically and radiographically, patients who will meet the eligibility criteria will be randomized. The standardized operating procedure of regenerative therapy requires two treatment visits. During the first appointment, infection is controlled and inflammation is relieved. Regenerative procedure and revascularization are accomplished during the second appointment. At the first visit, perioperative CBCT will be taken, access cavity with full mechanical preparation will be accomplished followed by application of double biotics paste for 3 weeks.

At the second appointment the intra-canal medicaments will be removed then 10 ml of blood of whole venous blood will be drawn from the patient's forearm and transferred into two plain plastic test tubes without an anticoagulant and will centrifuge immediately u at 700 rpm for 3 minutes then liquid platelet rich fibrin layer will be taken with plastic syringe and according to the group of the patient that will be assigned, the patient will receive either the iprf alone or to be mix with Vitamin C and injected inside the canal. Collagen membrane will be placed over the iprf or iprf with Vitamin C then the tooth will be restored with resin filling material, the patients will be followed every 3 months for 1 year, at every follow up periapical radiograph will be taken with standardized bite block and after 1 year CBCT will aslo be taken with same parameter of the perioperative one t be compared and asses the reduction of the periapical lesions

ELIGIBILITY:
Inclusion Criteria: Patients were enrolled to the present study if they fulfilled the inclusion criteria of being fit and healthy (ASA I and II).

* Adults with an age range of 18-45 years old, with no sex predication.
* Patients diagnosed with pulp necrosis in mature maxillary or mandibular anterior teeth with negative response to both cold and electrical pulp testing.
* Associated with or without swelling /sinus tract.
* Has radiographic evidence of periapical radiolucency

Exclusion Criteria: Patients with medically compromised conditions (ASA III and IV).

* Patients who are allergic to the drugs or pharmaceuticals used in the trial (mainly ciprofloxacin or metronidazole).
* Patients with presence of periodontal pockets, pathological mobility, ankyloses, root fracture.
* Patients with non-restorable teeth, teeth with pulp space needed for post cementation.
* Teeth with previous root canal treatment, teeth with developmental anomalies, and teeth with external or internal resorption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adults with an age range of 18-45 years old
Enrollment: 28 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Healing of periapical lesion | 1 year follow up
  Healing of periapical lesion will be assessed clinically normalcy including incidence of pain on percussion, swelling and sinus tract , aslo will be assed 2 dimensionally and 3 dimensionally using CBCT

SECONDARY OUTCOMES:
postoperative pain | 1 week
  postoperative pain will be assessed at 6, 12, 24, 48,72 hours and 1 week from the second visit using numerical pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Wesam Osama, assistant lecturer, Principal Investigator — Cairo University
Locations (1):
- Facility of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] 1-Tervit, C. et al. (2009) 'Proportion of Healed Teeth With Apical Periodontitis Medicated With Two Percent Chlorhexidine Gluconate Liquid: A Case-Series Study', Journal of Endodontics, 35(9), pp. 1182-1185. 2- Trope, M. (2003) The vital tooth-its importance in the study and practice of endodontics. Endod Topics 2003; 5:1-1. 3- Kim, S.G. et al. (2018) 'Regenerative endodontics: a comprehensive review', International Endodontic Journal. Blackwell Publishing Ltd, pp. 1367-1388. 4- Adnan, S. and Ullah, R. (2018) 'Top-cited Articles in Regenerative Endodontics: A Bibliometric Analysis', Journal of Endodontics. Elsevier Inc., pp. 1650-1664. 5- Kahler, B. and Lin, L.M. (2017) 'A REVIEW OF REGENERATIVE ENDODONTICS: CURRENT PROTOCOLS AND FUTURE DIRECTIONS', Journal of Istanbul University Faculty of Dentistry, 51(0). 6- Ibrahim, lamiaa, tawfik, mohamed and abu naeem, fatma (2021) "Evaluation of The Periapical Healing Following Pulp Revascularization Using Injectable PRF VS nonsurgical Root Canal Treatment in Mature Permanent Teeth with periapical periodontitis. A Clinical Study," Egyptian Dental Journal, 67(3), pp. 2663-2672.